## **Statistical Analysis Plan**

Shared Decision-Making: Implementing the AFib 2gether<sup>TM</sup> Mobile App

NCT #: NCT04118270

Date of document: 04/03/2020

For objective 1 regarding usability, we will calculate a composite score for both patients and providers. We will then norm this score to range from 0-100. If these norm scores fall along a normal distribution, we will calculate means and standard deviation for usability. Otherwise, we will group responses into categories and calculate frequencies. We will also calculate perceived usefulness for patients and providers and examine their distribution as we did for usability. In addition, we will record timing for each of the components of the shared decision-making encounter. We will review the distribution of time required for each activity. If they fall along a normal distribution, we will calculate means; otherwise, we will group into categories and calculate frequencies. We will then examine for trends in the association between certain patient factors such as age, gender, race, and income with the mobile app rating scale

For objective 2, to assess the association of provider knowledge of and, separately, confidence in modern AF management, we will examine each item in the Pfizer survey for consistency using factor analysis as well as our own expertise. If there are 1 or 2 factors that can summarize these responses, we will measure the association between a one category shift in knowledge or confidence and mean provider usability, mean provider perceived usefulness, and time-based feasibility.

For objective 3, we will track study patients' switch to AC using the EHR. More specifically we will calculate the frequency of patients starting anticoagulation up to six months after the shared decision-making visit.